CLINICAL TRIAL: NCT04532424
Title: Transcranial Magnetic Stimulation for Restricted and Repetitive Behavior in ASD
Acronym: TMS for ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-57738
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Autism; Asperger Syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of 2 groups based on the presentation of restricted and repetitive behavior.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Targeting insistence on sameness (Experimental)
  Interventions: Device: Transcranial magnetic stimulation
- Targeting stereotyped motor behaviors (Experimental)
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Non-invasive brain stimulation technique that is FDA-approved for the treatment of refractory depression, OCD and migraine.

SUMMARY:
Investigating the efficacy of a form of TMS called theta-burst stimulation for restricted and repetitive behavior in ASD.

ELIGIBILITY:
Inclusion criteria.

1. Diagnosis of Autism Spectrum Disorder (ASD)
2. Meet criteria for Autism Spectrum Disorder (ASD) on clinical assessments (ADOS-2 or CARS if conducted remotely & ADI-R)
3. Aged between 12-45 years old
4. Have a reliable informant who can complete relevant questionnaires
5. Have DARB scores which indicate high levels (50% or above) of RRB on one of the following domains: Insistence on Sameness, Obsessive Compulsive Behaviors, and Unusual Interests

Exclusion criteria.

1. Any contraindications for TMS e.g. history of seizures other than clear substance-induced/fever-induced seizures with neurologist note or normal clean EEG and no seizure in at least 12 months prior to enrollment.
2. Pregnancy.
3. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
4. Active substance use (<1 week) or intoxication verified by toxicology screen--of cocaine, amphetamines, benzodiazepines.
5. Showing symptoms of withdrawal from alcohol or benzodiazepines.
6. DSM-5 diagnosis of bipolar disorder or a psychotic disorder e.g. schizophrenia.
7. Significant sensory impairments such as blindness or deafness.
8. Current severe insomnia (must sleep a minimum of 4 hours the night before stimulation).
9. Not willing to cooperate with the TMS procedures.
10. Currently taking Clozapine or another medication that the PI determines increases the risk of TMS or may disrupt the efficacy.
11. A motor threshold that is too high to allow safe/tolerable treatment.
12. Conditions that increase the risk for COVID-19 (in accordance with university guidelines).

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Repetitive Behavior Scale-Revised (RBS-R) | Up to one month post-treatment
  44-item parent-report questionnaire to measure restricted and repetitive behavior in ASD. We predict that each TMS target will selectively reduce the subscale being targeted.

SECONDARY OUTCOMES:
Set-shifting performance (Dimensional Change Card Sort Test score) | Baseline & immediately after treatment
  The Dimensional Change Card Sort Test one of the cognitive measures from the NIH toolbox. These measures are administered on an iPad. The test takes 4 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barahona-Correa JB, Velosa A, Chainho A, Lopes R, Oliveira-Maia AJ. Repetitive Transcranial Magnetic Stimulation for Treatment of Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. Front Integr Neurosci. 2018 Jul 9;12:27. doi: 10.3389/fnint.2018.00027. eCollection 2018. PMID 30038561
- [Background] Oberman LM, Rotenberg A, Pascual-Leone A. Use of transcranial magnetic stimulation in autism spectrum disorders. J Autism Dev Disord. 2015 Feb;45(2):524-36. doi: 10.1007/s10803-013-1960-2. PMID 24127165